CLINICAL TRIAL: NCT03921073
Title: A Phase II Study of Talimogene Laherparepvec (T-VEC) in the Treatment of Locally Advanced Cutaneous Angiosarcoma
Brief Title: Study of T-VEC in Locally Advanced Cutaneous Angiosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Terminated Funding
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19878
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Angiosarcoma of Skin
Keywords: Cutaneous; Angiosarcoma; Skin
MeSH Terms: conditions — Hemangiosarcoma | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intralesional injection of T-VEC (Experimental): Participants will undergo intralesional injections of up to 4 cc of 10^6 plaque-forming units (PFU)/mL of T-VEC. Dose is dependent on the diameter of the lesions to be injected (volume injected is related to diameter of lesion(s) at time point 0). Three weeks later and every other week thereafter, the participants will be injected with up to 4 cc of 10^8 PFU/mL, with dose dependent on the diameter of the lesion(s) to be injected. Participants may be treated for up to 12 months.
  Interventions: Drug: T-VEC

INTERVENTIONS:
Drug: T-VEC — Participants will receive intralesional injections of T-VEC of up to 4cc. Dosing of T-VEC is dependent of the size of the lesion.

SUMMARY:
This is a single-arm study evaluating the efficacy of injecting Talimogene Laherparepvec T-VEC into Cutaneous Angiosarcoma tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed CA without visceral or CNS metastases, with resection deemed of no benefit by technical or oncologic principles, and have progressed on at least one line of systemic therapy
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded by digital photography) as >6 mm with calipers or a ruler.
* Eastern Cooperative Oncology Group performance status 0-1 (Karnofsky >70%).
* Participants must have normal organ and marrow function as defined below:
* Hematological
* Absolute neutrophil count > 1500/mm3 (1.5x109/L)
* Platelet count >75,000/mm3 (7.5x109/L)
* Hemoglobin >8 g/dL (without need for hematopoietic growth factor or transfusion support)
* Renal
* Serum creatinine ≤1.5 x upper limit of normal (ULN), OR 24-hour creatinine clearance >60 mL/min for subject with creatinine levels > 1.5 x ULN. (Note: Creatinine clearance need not be determined if the baseline serum creatinine is ≤1.5 x ULN. . Creatinine clearance should be determined per institutional standard).
* Hepatic
* Serum bilirubin ≤1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN
* Aspartate aminotransferase (AST) ≤2.5 x ULN OR <5 x ULN, if liver metastases present and injection does not involve a visceral lesion
* Alanine aminotransferase (ALT) ≤2.5 x ULN OR <5 x ULN, if liver metastases present and injection does not involve a visceral lesion
* Coagulation
* International normalization ratio (INR) or prothrombin time (PT) ≤1.5 x ULN, unless the subject is receiving anticoagulant therapy, in which case PT and partial thromboplastin time (PTT)/ activated PTT (aPTT) must be within therapeutic range of intended use of anticoagulants.
* PTT or aPTT ≤1.5 x ULN, unless the subject is receiving anticoagulant therapy as long as PT and PTT/aPTT is within therapeutic range of intended use of anticoagulants.- Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Exclusion Criteria:

* Participants with a second active malignancy, exceptions are localized non-melanoma skin cancers or in situ carcinoma
* Participants receiving any other investigational agents
* Participants with tumor(s) in direct contact or encasing a major blood vessel, those with ulceration and/or fungation onto the skin surface, and those with history of re-irradiation or prior lymph node neck dissection to a field involving the carotid arteries
* History or evidence of active autoimmune disease that requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Evidence of clinically significant immunosuppression such as the following:
* Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease.
* concurrent opportunistic infection.
* receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrollment.
* Active herpetic skin lesions or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis).
* Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.
* Previous treatment with talimogene laherparepvec or any other oncolytic virus.
* Prior therapy with tumor vaccine.
* Received live vaccine within 28 days prior to enrollment.
* Prior immunosuppressive, chemotherapy, radiotherapy (in which the field encompassed a planned injection site), biological cancer therapy, or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment.
* Prior radiotherapy in which the field does not overlap the injection sites or non-immunosuppressive targeted therapy within 14 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 14 days prior to enrollment
* Currently receiving treatment with another investigational device or drug study, or < 28 days since ending treatment with another investigational device or drug study(s).
* Other investigational procedures while participating in this study are excluded.
* Known to have acute or chronic active hepatitis B infection, hepatitis C infection, or human immunodeficiency virus (HIV) infection.
* History of other malignancy within the past 5 years with the following exceptions: adequately treated non melanoma skin cancer, cervical carcinoma in situ, breast ductal carcinoma in situ, or prostatic intraepithelial neoplasia without evidence of disease at the time of enrollment
* Participant has known sensitivity to talimogene laherparepvec or any of its components to be administered during dosing.
* Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of talimogene laherparepvec.
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec.
* Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec.
* Participants who are unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or infants under the age of 3 months, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mullinax, MD,, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intralesional Injection of T-VEC
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intralesional Injection of T-VEC
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is defined as the proportion of patients who demonstrate complete or partial responses in injected lesions per modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria appropriate for cutaneous neoplasms (ORR=complete response + partial response).
Time Frame: at 24 Weeks
Population: Data not collected. 0 participants analyzed. Study terminated early.
Arm/Group | Intralesional Injection of T-VEC
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response
Description: Response duration will be measured from the time of initial partial response or complete response until documented progression.
  The duration of overall response is measured from the time measurement criteria are met for Complete Response or Partial Response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: at 4 weeks
Population: Data not collected. 0 participants analyzed. Study terminated early.
Arm/Group | Intralesional Injection of T-VEC
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the period of time from the first injection to progression of disease or appearance of new cutaneous angiosarcomas that were not present at the time of study entry
Time Frame: up to 2 years
Population: Data not collected. 0 participants analyzed. Study terminated early.
Arm/Group | Intralesional Injection of T-VEC
Number analyzed (Participants) | 0

4. Secondary Outcome: Complete Response Rate
Description: Complete response rate is defined as the proportion of participants that have lesions with complete clinical regression
Time Frame: Baseline to 2 years
Population: Data not collected. 0 participants analyzed. Study terminated early.
Arm/Group | Intralesional Injection of T-VEC
Number analyzed (Participants) | 0

5. Secondary Outcome: T-VEC Treated Tumors Requiring Surgical Resection
Description: Measuring the rate of participants requiring surgical resection of T-VEC treated lesions
Time Frame: Baseline to 2 years
Population: Data not collected. 0 participants analyzed. Study terminated early.
Arm/Group | Intralesional Injection of T-VEC
Number analyzed (Participants) | 0

6. Secondary Outcome: Analyses of Immune Infiltration Within Resected Tumor Specimens
Description: Measuring the degree of immune infiltration in surgically resected T-VEC treated tumors
Time Frame: Baseline to 2 years
Population: Data not collected. 0 participants analyzed. Study terminated early.
Arm/Group | Intralesional Injection of T-VEC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected from date on treatment to 30 days after off treatment date, for an average of 9 months
Description: No anticipated or unanticipated serious adverse events happened to participants on trial.
Arm/Group | Intralesional Injection of T-VEC
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intralesional Injection of T-VEC (N=5)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2)
Periorbital edema (Eye disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 3 (7)
Flu like symptoms (General disorders) | 3 (30)
Injection site pain (General disorders) | 3 (4)
Pain (General disorders) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scalp (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03921073/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT03921073/ICF_002.pdf